CLINICAL TRIAL: NCT03075228
Title: DUPLO Study: Comparison of the Microbial Composition of the Upper Gastrointestinal Tract in Lean and Obese Subjects
Brief Title: Comparison of the Microbial Composition in Lean and Obese Subjects
Acronym: DUPLO
Status: Terminated | Type: Observational
Why Stopped: Low recruitment rate; high proportion of screening failures.
Sponsor: NIZO Food Research (Other)
Collaborators: Danisco Sweeteners Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: NL 59327.081.16
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: microbiota; small intestine; metabolic disease
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, fecal samples, small intestinal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean subjects: Lean is defined as having a BMI of 19-23 kg/m2, waist circumference <80 cm and fasting glucose levels <6.1 mmol/L.
  Interventions: Device: IntelliCap
- Obese subjects: Obese is defined as having a BMI of 30-35 kg/m2, waist circumference >88 cm and fasting glucose levels >=6.1 and <7.5 mmol/L
  Interventions: Device: IntelliCap

INTERVENTIONS:
Device: IntelliCap — Sampling of the small intestine using a samling capsule.

SUMMARY:
Rationale: The microbial composition in the small intestine (SI) differs largely from the composition in feces. Many physiological processes related to health, such as immunoregulation and metabolic programming, mainly take place in the SI. Therefore, the SI, from a microbiota perspective, is as relevant as the large intestine. There are indications that microbiota composition is different in lean and obese subjects, and is related to insulin resistance. However, these indications are mainly based on the analysis of fecal samples. Therefore, analysis of the microbiota composition in the more proximal part of the gastrointestinal (GI) tract may provide new insights into the microbial species that are involved or related to metabolic homeostasis at that location. The IntelliCap® CR system offers a minimally invasive tool that is able to collect reliable samples in the SI, as was shown by NIZO in a clinical validation study. The main aim of the current study is to explore and compare the upper GI microbiota composition in lean and obese subjects, in order to generate new leads for development of products that may target the upper GI microbiota community or specific species thereof, which may impact the maintenance of metabolic homeostasis. This may provide new opportunities for the treatment, reduction or prevention of overweight and/or obesity or insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age: 25-50y;
* Lean: BMI 19-23 kg/m2, waist circumference <80 cm, and fasting glucose <6.1 mmol/L; Obese: BMI 30-35 kg/m2, waist circumference >88 cm, and fasting glucose >=6.1 and <7.5 mmol/L;
* Healthy as assessed by the NIZO lifestyle and health questionnaire ("Verklaring leefgewoonten en gezondheid");
* Healthy as assessed by results of the pre-study safety laboratory tests (clinical chemistry: liver/kidney function etc);
* Regular and normal Dutch eating habits as assessed by the NIZO lifestyle and health questionnaire (3 main meals per day);
* Regular bowel movement (defecation on average once a day, at least 4 times/week).

Exclusion Criteria:

* Participation in any clinical trial with oral, intravenous or inhalatory administration of any substances during 90 days before study start;
* History or presence of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study:

  * type 1 or type 2 diabetes;
  * gastrointestinal disease;
  * bariatric surgery;
  * cardiovascular disease, liver or renal failure or disease of the thyroid gland, cancer;
  * infectious disease, history of chronic active inflammatory disorders or food allergy;
* Use of antibiotics during the one (1) year prior to study start; #
* Constipation/infrequent bowel movement (defecation <4 times per week);
* Having diarrhea within 3 months prior to the study start (at least 3 loose stools per day);
* Use of laxatives, fiber supplements (e.g. lactulose, inulin), glucose lowering drugs, insulin, anti-obesity drugs, immunosuppressive drugs (e.g. systemic corticosteroids, cyclosporine, azathioprine, antibodies) during the three (3) months prior to study start;
* Use of temporary or irregular medication for diabetes, dyslipidemia or hypertension;
* Use of any prescribed or non-prescribed medication (other than paracetamol) including antacids, H2 receptor antagonists, proton pump inhibitors, analgesics, herbal remedies or anti-inflammatory drugs (e.g. NSAIDs) during the three (3) weeks prior to study start;
* Use of probiotics or prebiotics during the three (3) months prior to study start;
* Mental status that is incompatible with the proper conduct of the study;
* Presence of swallowing or passage disorder;
* Carrying a pacemaker or any other (implanted) medical electronic device;
* Scheduled for an MRI scan during the study period;
* Not willing to have an X-ray if the capsule is not recovered from the faeces;
* Alcohol consumption > 15 units/week and >3/day. In case of less alcohol consumption: not willing to stop during the study;
* Drug abuse, and not willing/able to stop this during the study;
* Heavy exercise or sports training > 10 hours/week;
* Smoking;
* Active or recent participation in a weight loss program including weight change (increase or loss) of >3 kg during the last three (3) months;
* Reported unexplained weight loss or weight gain of > 5 kg in the year prior to pre-study screening;
* Reported slimming or medically prescribed diet;
* Reported special diets;
* Pregnant or planning to become pregnant during the study, breastfeeding ;
* Postmenopausal women on unstable hormone replacement therapy.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ten (10) apparently healthy lean female subjects, as well as ten (10) apparently healthy obese female subjects, all aged 25-50y, will be recruited locally/regionally from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Microbiota composition | 3 days after consuming a fully controlled western style diet
  Relative abundance of microbiota species (% of total) in the small intestine in lean vs obese subjects

SECONDARY OUTCOMES:
Total bacterial count | 3 days after consuming a fully controlled western style diet
  Total bacterial count measured by qPCR in the small intestinal samples in lean vs obese subjects
Cytokine levels | 3 days after consuming a fully controlled western style diet
  Cytokines levels in blood in relation to microbiota composition in lean vs obese subjects
Metabolic markers | 3 days after consuming a fully controlled western style diet
  Glucose, insulin and cholesterol levels in blood in relation to microbiota composition in lean vs obese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Els van Hoffen, PhD, Principal Investigator — NIZO food research BV
Locations (1):
- NIZO food research BV, Ede, Netherlands

IPD SHARING:
Plan to Share IPD: No